CLINICAL TRIAL: NCT04900532
Title: Effects of Supplementation With Tocotrienol on Inflammation, Oxidative Stress and Microbiota of Chronic Kidney Disease Patients
Brief Title: Effects of Supplementation With Tocotrienol on Chronic Kidney Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Collaborators: Wayne State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: Denise Mafra
Record Dates: First submitted 2020-12-04; First posted 2021-05-25 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Chronic Kidney Diseases; Hemodialysis; Microbiota; Oxidative Stress; Inflammation
MeSH Terms: conditions — Renal Insufficiency, Chronic; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effects of supplementation with tocotrienol on chronic kidney disease patients (Experimental): Administration of tocotrienol-rich-fraction (TRF) capsules, containing 360mg of tocotrienol and 80mg of tocopherol twice a day for six months.
  Interventions: Dietary Supplement: Tocotrienol rich fraction
- Effects of supplementation with tocotrienol on lipid profile of chronic kidney disease patients (Placebo Comparator): Administration of placebo containing 0,96mg of tocotrienol and 1,76mg of tocopherol twice a day for three months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Tocotrienol rich fraction — Supplementation with a Vitamin E compound.
  Arms: Effects of supplementation with tocotrienol on chronic kidney disease patients
Dietary Supplement: Placebo — Administration of placebo containing 0,96mg of tocotrienol and 1,76mg of tocopherol twice a day for three months.
  Arms: Effects of supplementation with tocotrienol on lipid profile of chronic kidney disease patients

SUMMARY:
The objective of this study is to evaluate the supplementation with tocotrienol, a vitamin E compound on inflammation, oxidative stress, and microbiota on Chronic Kidney Disease patients.

DETAILED DESCRIPTION:
In Chronic Kidney Disease (CKD), inflammation and oxidative stress are common statuses, which are aggravated by renal replacement therapy such as hemodialysis. Currently, intestinal microbiota imbalance has been associated with both inflammation and oxidative stress. In this regard, strategies in the management of this framework are necessary. It has been observed that vitamin E plays an important role in the modulation of transcription factors involved in inflammation such as NF-kB and Nrf2, acting on cell membrane protection and tissue recovery. Its benefits have been proven both in renal and intestinal health, however, studies analyzing the vitamin E supplementation in the modulation of intestinal microbiota with consequent effect on CKD and its reflexes are scarce. Thus, the current randomized, double-blind, placebo-controlled study will evaluate the effects of vitamin E supplementation on the modulation of the expression of nuclear cytokine (NF-kB e Nrf2), activators and inhibitors, as well as, on inflammation and oxidative stress and on the modulation of the intestinal microbiota in patients CKD.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease
* Aged from 18 to 60 years
* Must be able to swallow capsules

Exclusion Criteria:

* Pregnant patients
* Smokers
* Using antibiotics in the last 3 months
* Using antioxidant supplements in the last 3 months
* Usual intake Autoimmune
* Hemodialysis started less than 6 months for hemodialysis patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in antioxidants and anti-inflammatory biomarkers | 4 weeks
  Get blood samples to evaluate the supplementation effects in antioxidants biomarkers- nuclear receptor factor 2 (Nrf2), glutathioneperoxidase (GPx), heme oxygenase-1 (HO-1).
  glutathione peroxidase (GPx), heme oxygenase-1 (HO-1) and microbiota composition from patients feces DNA uremic toxins

SECONDARY OUTCOMES:
Change in inflammatory biomarkers | 4 weeks
  Get blood samples to evaluate the supplementation effects in inflammatory biomarkers- factor nuclear kappa B (NFkB), interleukin 6 (IL-6), tumor necrosis factor alpha (TNF-alpha).

CONTACTS AND LOCATIONS:
Locations (1):
- Denise Mafra, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Trugilho L, Alvarenga L, Cardozo L, Paiva B, Brito J, Barboza I, Almeida J, Dos Anjos J, Khosla P, Ribeiro-Alves M, Mafra D. Effects of Tocotrienol on Cardiovascular Risk Markers in Patients With Chronic Kidney Disease: A Randomized Controlled Trial. J Nutr Metab. 2025 Jan 13;2025:8482883. doi: 10.1155/jnme/8482883. eCollection 2025. PMID 39840146